CLINICAL TRIAL: NCT01739907
Title: Iron-fortified Flavoured Skimmed Milk With or Without Vitamin D in Iron Deficient Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, M Pilar Vaquero, Scientific researcher, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AGL2009-11437
Record Dates: First submitted 2012-11-20; First posted 2012-12-04 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2012-11

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; Menstruating women; Vitamin D; Functional food
MeSH Terms: conditions — Iron Deficiencies | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron-fortified dairy product (Experimental): Consumption of an iron-fortified flavoured skimmed milk as part of the usual diet
  Interventions: Other: Iron fortified flavoured skimmed milk with or without vitamin D in iron deficient women
- Iron and vitamin D dairy product (Experimental): Consumption of an iron and vitamin D fortified flavoured skimmed milk as part of the usual diet
  Interventions: Other: Iron fortified flavoured skimmed milk with or without vitamin D in iron deficient women

INTERVENTIONS:
Other: Iron fortified flavoured skimmed milk with or without vitamin D in iron deficient women

SUMMARY:
Iron deficiency and vitamin D deficiencies are common in menstruating women. The present assay studied the influence of the consumption of a flavoured skimmed milk with iron (iron pyrophosphate) or with iron and vitamin D3 in iron deficient women on:

* Iron metabolism
* Biomarkers of bone remodelling
* Cardiovascular risk indexes

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker or smokers of ≤ 3 cigarettes/day
* Non-pregnant
* non-breast-feeding
* Serum ferritin <30ng/mL
* Haemoglobin ≥11g/dL

Exclusion Criteria:

* Amenorrhea
* Menopause
* Any known health problems likely to influence iron status including iron-metabolism-related diseases (iron deficiency anaemia, thalassaemia, haemochromatosis)
* Chronic gastric diseases (inflammatory bowel disease, Crohn disease, gastric ulcers, celiac disease, hemorrhagic diseases)
* Renal disease or allergy to some of the components of the assay diary product.
* Blood donors
* Have regularly consumed iron or ascorbic acid supplements within the four months prior to participating in the intervention.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ferritin changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)

SECONDARY OUTCOMES:
Haemoglobin changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Total erythrocytes changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Haematocrit changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Mean corpuscular volume changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Red blood cell distribution width changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Serum iron changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Serum transferrin changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Transferrin saturation changes over 16 weeks | 16 weeks (Measures at 0, 4, 8, 12 and 16 weeks)
Soluble transferrin receptor changes over 16 weeks | 16 weeks (Measures at 0, 8, and 16 weeks)
25-hydroxyvitamin D changes over 16 weeks | 16 weeks (Measures at 0, 8, and 16 weeks)
Procollagen type 1 N-terminal propeptide (P1NP) changes over 16 weeks | 16 weeks (measures at 0, 8 and 16 weeks)
Cross-linked N-telopeptides of type I collagen (NTX) changes over 16 weeks | 16 weeks (measures at 0, 8 and 16 weeks
Parathormone (PTH) changes over 16 weeks | 16 weeks (measures at 0, 8 and 16 weeks
Total cholesterol changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks
LDL-cholesterol changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)
HDL-cholesterol changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)
Triglycerides changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)
Systolic blood pressure changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)
Diastolic blood pressure changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)
glucose changes over 16 weeks | 16 weeks (Measures at 0, 8 and 16 weeks)

REFERENCES:
- [Background] Blanco-Rojo R, Toxqui L, Lopez-Parra AM, Baeza-Richer C, Perez-Granados AM, Arroyo-Pardo E, Vaquero MP. Influence of diet, menstruation and genetic factors on iron status: a cross-sectional study in Spanish women of childbearing age. Int J Mol Sci. 2014 Mar 6;15(3):4077-87. doi: 10.3390/ijms15034077. PMID 24663082
- [Background] Wright I, Blanco-Rojo R, Fernandez MC, Toxqui L, Moreno G, Perez-Granados AM, de la Piedra C, Remacha AF, Vaquero MP. Bone remodelling is reduced by recovery from iron-deficiency anaemia in premenopausal women. J Physiol Biochem. 2013 Dec;69(4):889-96. doi: 10.1007/s13105-013-0266-3. Epub 2013 Jun 28. PMID 23813442
- [Result] Toxqui L, Perez-Granados AM, Blanco-Rojo R, Wright I, Gonzalez-Vizcayno C, Vaquero MP. Effects of an iron or iron and vitamin D-fortified flavored skim milk on iron metabolism: a randomized controlled double-blind trial in iron-deficient women. J Am Coll Nutr. 2013;32(5):312-20. doi: 10.1080/07315724.2013.826116. PMID 24219374
- [Result] Toxqui L, Perez-Granados AM, Blanco-Rojo R, Wright I, de la Piedra C, Vaquero MP. Low iron status as a factor of increased bone resorption and effects of an iron and vitamin D-fortified skimmed milk on bone remodelling in young Spanish women. Eur J Nutr. 2014;53(2):441-8. doi: 10.1007/s00394-013-0544-4. Epub 2013 Jun 16. PMID 23771807
- [Result] Toxqui L, Blanco-Rojo R, Wright I, Perez-Granados AM, Vaquero MP. Changes in blood pressure and lipid levels in young women consuming a vitamin D-fortified skimmed milk: a randomised controlled trial. Nutrients. 2013 Dec 5;5(12):4966-77. doi: 10.3390/nu5124966. PMID 24317556
- [Result] Toxqui L, Perez-Granados AM, Blanco-Rojo R, Wright I, Vaquero MP. A simple and feasible questionnaire to estimate menstrual blood loss: relationship with hematological and gynecological parameters in young women. BMC Womens Health. 2014 May 30;14:71. doi: 10.1186/1472-6874-14-71. PMID 24886470